CLINICAL TRIAL: NCT06822452
Title: Prospective Comparative Study Evaluating the Early Complications of Robot-assisted Radical Prostatectomy Performed as an Outpatient Versus an Inpatient Procedure.
Acronym: PROSTAMBU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PROSTAMBU; 2024-A01745-42 (Other: ID-RCB)
Record Dates: First submitted 2025-01-31; First posted 2025-02-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer Surgery; Ambulatory Care; Outpatient Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Outpatient procedure (Experimental)
  Interventions: Procedure: radical prostatectomy
- Inpatient procedure (Active Comparator)
  Interventions: Procedure: radical prostatectomy

INTERVENTIONS:
Procedure: radical prostatectomy — Robot-assisted

SUMMARY:
The goal of this clinical trial is to demonstrate that outpatient management for robotic-assisted radical prostatectomy is not inferior to inpatient management in terms of the occurrence of early post-operative complications.

Researchers will compare outpatient robot-assisted radical prostatectomy to inpatient procedure.

Participants will:

* Visit the clinic after the operation once at 45 days, 6 months and once a year for up to 5 years for check-ups and tests.
* Answer survey questions about urinary and erectil functions, stress and anxiety, satisfaction, quality of life for 6 months
* Keep a diary to record procedures and treatments related to the care provided

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 and over
* Patient with prostate cancer for which the multidisciplinary meeting has proposed radical prostatectomy as a therapeutic option (with or without lymphadenectomy)
* Patient eligible for outpatient treatment :

  1. The patient undertakes to comply with all medical instructions given during surgical consultations and the anaesthetic consultation.
  2. The patient has access to personal transport allowing, if necessary, return to the facility or another approved facility (transport time and distance from the facility are not exclusion factors)
  3. The patient has access to telephone communication facilities.
  4. The patient undertakes not to drive a vehicle and to be accompanied on his return home and for the next 24 hours by a responsible person who will be familiar with the monitoring instructions.
  5. The patient plans to remain in hospital overnight if this is deemed necessary by the department's doctors (operator and anaesthetist). The patient accepts this mode of care and its constraints.
* Participant affiliated to or benefiting from a social security scheme
* The participant has been informed and has given his/her free, informed and written consent (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patient already treated for prostatic carcinoma with brachytherapy, radiotherapy or focal therapy
* Patient participating in ongoing research or in a period of exclusion at the time of inclusion
* Refusal or inability to comply with the study protocol for any reason whatsoever
* Protected participant: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2027-01-07 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Early complication of robot-assisted prostatectomy | From the day of surgery to 8 days post-operative
  The occurrence (yes/no) of at least one early complication of robot-assisted prostatectomy.
  The early clinical complications expected are :
  * Bleeding from trocar incision scars or surgical excision scars
  * Urinary leakage around the catheter
  * Retention due to bladder catheter clotting
  * Loss of bladder catheter
  * Signs of internal haemorrhage (within 24 hours)
  * Signs of biological deglobulation
  * Intestinal obstruction syndrome
  * Signs of urinary fistula
  * Infectious signs : fever > 38°, chills
  * Thromboembolicaccidents
  * Nosocomial infections
  * Falls

SECONDARY OUTCOMES:
Conversion rate from outpatient to full hospitalisation (Outpatient failure rate) | Day of surgery
  Patients treated on an outpatient basis for whom full hospitalisation is indicated on the day of surgery, as decided by the medical team.
Rate of cancellation of outpatient treatment by the patient or his private environment | From enrollment to the day of surgery
  Patients included in the study refusing outpatient care up to the day of surgery (before or after surgery) for whatever reason
Rate of patients readmitted to hospital, either as emergencies or in the department | From hospital discharge to 8 days post-operative.
  Patients readmitted to hospital (yes/no), emergency or inpatient department
Association of each early complication with treatment (outpatient or inpatient) | From hospitalisation discharge to 8 days post-operative
  Early complication of robot-assisted prostatectomy
Rate of patients having had at least one complication secondary to surgery | From 8 days to 45 days post-operative
  Patients who had at least one complication secondary to surgery.
  The expected complications secondary to surgery are:
  * Admission to emergency care
  * Re-hospitalization
  * Occlusions
  * Healing problems
  * Perineal hematoma
  * Urinary infections
  * Lymphoceles
  * Thromboembolic accidents
  * Nosocomial infections
Rate of patients with at least one complication secondary to surgery | From 45 days to 6 months post-operative
  Patients who had at least one complication secondary to surgery.
Patient's pre-operative stress/anxiety levels | 3 days before surgery, day of surgery and 2 days post-operative
  The participant's stress/anxiety level is assessed at 3 days before surgery using the APAIS (Amsterdam Preoperative Anxiety and Information Scale) questionnaire validated in French (Moerman and al, 1996; Maurice-Szamburski and al, 2013), then with a Numerical Scale of stress/anxiety during preparation for the operating theatre in the care unit and at 2 days post-operative.
Patient satisfaction level | 2 days and 45 days post-operative
  Patient satisfaction is assessed using the overall satisfaction question in the e-SATIS questionnaire ("Overall, how would you rate the quality of your treatment/care in the department by the doctors/surgeons/nurses? Bad/Weak/Average/Good/Excellent) The patient's opinion (yes/no) is evaluated on whether, if the procedure were repeated, the patient would accept it (yes/no) and whether it reassured him/her to go home in the evening /stay in hospital at night after the procedure.
Duration of surgery | Day of surgery
  Duration of surgery 'skin-to-skin' (incision until final stitch complete)
Blood loss | Day of surgery
  The level of blood loss is assessed by the quantity of blood recovered in the aspiration jar and the quantity from the drains minus the quantity perfused intraoperatively in ml.
Rate of patients who recovered continence and rate of patients who recovered urinary function after surgery | Baseline and 45 days post-operative
  Urinary continence is assessed by the response to question 5 of the EPIC-50 (Expanded Prostate Cancer Index Composite) when 0 to 1 pads are used during the day by the patient. Recovery of urinary function was assessed by the difference between the incontinence subscore of the EPIC-50 questionnaire at D45 and the value of the pre-operative score.
  The incontinence subscore include questions 1, 3, 4, 5 and 6a of the urinary function EPIC-50 questionnaire. The EPIC-50 is a validated questionnaire (Wei and al, 2000) and translated into French (Anota and al, 2016).
Evolution of urinary continence between 45 days and 6 months post-operatively and evolution of urinary function pre-operatively, at 45 days, at 6 months. | Baseline and 45 days, 6 months after surgery
  The evolution of continence and urinary function is established on the basis of the parameters defined previously (see Secondary Outcome Measure 12.)
Recovery of erectile function | Baseline and 6 months post-operative
  Erectile recovery is assessed using the IIEF-5 (International Index of Erectile Function) questionnaire (Rosen R and al, 1997; Dargis and al, 2013) ; erectile dysfunction is defined by an IIEF-5 score <10.
Oncological recurrence and retreatment | From 45 days to 5 years after surgery
  Recurrence is defined by a PSA (Prostate Specific Antigen) level >0.1ng/ml, the patient's re-treatment (yes/no), the type of re-treatment (hormone therapy / chemotherapy / radiotherapy).
Economic and social cost of patient care | From hospital discharge to 6 months post-operative
  The cost-utility ratio calculated on the basis of :
  - The costs of the homogeneous group of patients (GHM) for hospitalisation and the costs of the national care reference system (ENCC) for post-operative management, based on the patient's diary completed up to 6 months after the operation.
  The following direct medical costs will be estimated from a societal perspective with a time horizon of 6 months:
  * Medical transport, medical and non-medical consultations in town, complementary examinations and drugs: collected in the CRF of the study from the patient logbook and valued using current tariffs.
  * The QALY, a unit for measuring life expectancy weighted by health-related quality of life, calculated on the basis of the utility derived from the EQ-5D-5L quality of life questionnaire completed by the patient at D0, D45 and 6 months after surgery.

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Clinique Rhône Durance, Avignon
  - Clinique St Vincent, Besançon
  - Clinique St Augustin, Bordeaux
  - Polyclinique Médipôle St-Roch, Cabestany
  - Polyclinique du Parc, Caen
  - Pole Sante Sud-CMCM, Le Mans
  - Hôpital Privé Nancy Lorraine, Nancy
  - Polyclinique Les Fleurs, Ollioules
  - Polyclinique Santé Atlantique, Saint-Herblain
  - Clinique Belledonne, Saint-Martin-d'Hères
  - Centre clinical, Soyaux
  - Hôpital Privé Océane, Vannes

IPD SHARING:
Plan to Share IPD: No